CLINICAL TRIAL: NCT01400308
Title: Clinical Trial to Compare the Effectiveness of Two Protocols for Corporal Decolonization in Patients Colonized by MRSA (Methicillin Resistant Staphylococcus Aureus)
Brief Title: Effectiveness of Two Protocols for Corporal Decolonization in Patients Colonized by Methicillin Resistant Staphylococcus Aureus (MRSA)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The differences seen between treatments led to recalculation of the sample, unattainable in a reasonable time
Sponsor: B. Braun Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPM-G-H-0903
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: MRSA - Methicillin Resistant Staphylococcus Aureus Infection; MRSA Colonization
Keywords: Methicillin Resistant Staphylococcus Aureus colonization.; Methicillin Resistant Staphylococcus Aureus infection.
MeSH Terms: interventions — Mupirocin; Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine + Mupirocin (Active Comparator): Will be treated with the protocol described in the "Consensus document and GEIH-SEIMC SEMPSPH" Version 31/10/07, as shown listed in Table 4. It is a protocol of 5 days (nasal mupirocin and chlorhexidine, potentially plus systemic antibiotics and 7 days).
  Interventions: Drug: Mupirocin + Chlorhexidin
- Prontoderm (Experimental): Will be treated with the protocol established for Prontoderm® for five days and eventually plus systemic antibiotics.
  Interventions: Device: Prontoderm MRSA Kit

INTERVENTIONS:
Drug: Mupirocin + Chlorhexidin — Treatment after protocol described in the "Consensus document and GEIH-SEIMC SEMPSPH" Version 31/10/07. It is a protocol of 5 days (nasal mupirocin and chlorhexidine, potentially plus systemic antibiotics and 7 days)
  Arms: Chlorhexidine + Mupirocin
Device: Prontoderm MRSA Kit — Treatment after protocol established for Prontoderm® for five days and eventually plus systemic antibiotics.
  Prontoderm® is a Class III medical device
  Arms: Prontoderm

SUMMARY:
Multicenter Clinical Trial, experimental, randomized and prospective study to determine the effectiveness of two protocols addressing the Corporal Decolonization in patients colonized by Methicillin Resistant Staphylococcus Aureus (MRSA).

PRIMARY END POINT The aim of this trial is to evaluate the effectiveness of the protocol Prontoderm® in the decolonization of MRSA patients, compared with the protocol of the "Consensus Document and GEIH-SEIMC SEMPSPH" (see attached extract from the document, Annex 7).

Prontoderm ® is a Class III Medical Device with CE mark owned by B.BRAUN Medical SA, and currently available in Spain for the same indications proposed in this trial.

DETAILED DESCRIPTION:
Design: Multicenter, experimental, randomized and prospective study. The patients were consecutively and alternately assigned to each comparison group. Randomization was assured by central randomization and the first patient to one of the groups and, from there, too centrally, back to each of the two groups.

Group A will be treated with the protocol described in the "Consensus document and GEIH-SEIMC SEMPSPH" Version 31/10/07, as shown listed in Table 4. It is a protocol of 5 days (nasal mupirocin and chlorhexidine, potentially plus systemic antibiotics and 7 days).

Group B will be treated with the protocol established for Prontoderm® for five days and eventually plus systemic antibiotics. Ensure the correct application of the treatments without interruption over the weekend indicated protocol.

Sample Calculation: The investigators propose an initial sample of 310 patients for a bilateral approach with a type I error α = 0.05 and β type II error of 20%.

Analysis:

Simple analysis and logistic regression (to adjust for risk factors, sources, concomitant therapy, etc) compared the frequency of decolonization of MRSA, according to sources.

Procedures: To collect information using a standardized form CRD in paper to all hospitals, indicating the parameters listed in this protocol and cultures to be done both baseline and monitoring cultures

DISEASE IN STUDY

This will be treated either or both of the following conditions:

MRSA Colonization: The presence of the organism in the flora of the patient, detected by positive culture for MRSA, and no diagnosis of infection.

MRSA infections: presence of the organism between the flora of the patient, detected by positive culture for MRSA, and the presence of MRSA infection diagnosed according to criteria EPINE 2009 (Annex 8).

ELIGIBILITY:
Inclusion Criteria:

- MRSA infected or colonized Patients

Exclusion Criteria:

Patients whose condition or treatment interferes with the proper implementation of the proposed protocols, such as:

* Patients admitted to the ICU
* Patients undergoing resuscitation
* Immobilized patients-avoiding their complete hygiene
* Patients carrying nasogastric tube
* Patients with tracheostomy and / or assisted mechanical ventilation
* Patients who are unable, neither they nor their representatives, to give valid informed consent.
* Patients whose discharged is planned before completing protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Decolonization of MRSA patients | Final treatment day + 4 (by second control sample)
  The aim of this trial is to evaluate the effectiveness of the protocol "Prontoderm ® in the decolonization of MRSA patients", compared with the protocol of the "Consensus Document and GEIH-SEIMC SEMPSPH" Prontoderm ® is a Class III Medical Device with CE mark owned by B.BRAUN Medical SA, and currently available in Spain and all over Europe for the same indications proposed in this trial.

SECONDARY OUTCOMES:
Percent of decolonization out of total by trained staff treated patients | Up to two years
  For both arms, determine the importance of staff training and the proper procedure in the application of hygiene measures, by comparing trial outcomes with same centre historical outcomes regarding MRSA decolonization
Quantitative (0-10 scale) and qualitative (open questions) measure of the usability of experimental and control products by users | The fifth, final day of treatment
  Measure of user satisfaction regarding the usability of the experimental product vs control, by self-administered questionnaire. The fifth and final day of treatment the staff fills out a questionnaire that includes questions about product usability
Quantitative (0-10 scale) and qualitative (open questions) measure of the acceptance of experimental and control products by staff | The fifth, final day of treatment
  Measure of user satisfaction regarding features of the experimental product vs control, by self-administered questionnaire. The fifth and final day of treatment the staff fills out a questionnaire that includes questions about products' features
Quantitative (0-10 scale) and qualitative (open questions) measure of the organoleptic features of experimental and control products by patients | The fifth, final day of treatment
  Measure of patient rating satisfaction regarding the organoleptic features of the experimental product vs control, by self-administered questionnaire.The fifth and final day of treatment the staff fills out a questionnaire that includes questions about product organoleptic features
Quantitative (0-10 scale) and qualitative (open questions) measure of the acceptance of experimental and control products by patient | The fifth, final day of treatment
  Measure of patients' satisfaction regarding features of the experimental product vs control product, by self-administered questionnaire. The fifth and final day of treatment the patient fills out a questionnaire that includes questions about product acceptance
Percent of decolonization in with Prontoderm® treated multiresistant colonizations decolonization for other multiresistant organisms (not MRSA) | After completation of treatment (5 days) two culture are done (2nd day and forth day after finishing) and colonizationd + resistances are mesured
  Rate effectiveness of Prontoderm® for other multiresistant organisms (such as Acinetobacter, Pseudomonas, Vancomycin Resistant Enterococcus , E. Coli, Klebsiella and other Enterobacteriaceae producing ESBL).
  In the pretreatment culture not only MRSA but also other of the above mentioned bacteria can appear. After finishing treatment, the decolonization of these other bacteria will be assessed (effectiveness of product)
Incidence and prevalence of multidrug resistant bacteria after experimental vs control treatment | After completation of treatment (5 days) two culture are done (2nd day and forth day after finishing) and colonizationd + resistances are mesured
  To assess the difference in the appearance of multidrug resistance between both arms
Delta (decrease or increase) in MRSA epidemiology (incidence, prevalence) for the centre comparing the years before trial and after trial | Up to two years
  Mesure of impact of the experimental protocol on the epidemiology by measuring the decrease or increase in MRSA epidemiology (incidence, prevalence) after applying the experimental protocol compared with historical figures from the center- in hospitals where there is a vigilance system for nosocomial infection
Assess the efficiency (economic impact) of the proposed protocol | Up to two years
  Costs of both (experimental and control) treatments will be compared, considering not only price of products, but other MRSA treatment related resources such as staff time, isolation days, etc, to assess the efficiency, economic impact, of the proposed protocol with Prontoderm®, compared with control treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Ortí, Dr., Principal Investigator — Responsible for Preventive Medicine Hospital Clínic Universitari de Valencia
Locations (4):
- Spain (4):
  - Hospital General Universitario de Elche., Elche, Valencia
  - Hospital Clínic Universitari de Valencia., Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia, Valencia
  - Hospital Universitari de Bellvitge, Barcelona